CLINICAL TRIAL: NCT04949737
Title: Prevalence of Helicobacter Pylori Infection and Gastric Cancer in the West Indies: Helico-MQ Interventional Study
Brief Title: Prevalence of Helicobacter Pylori Infection and Gastric Cancer in the West Indies
Acronym: Hélico-MQ
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH2_22; 2020-A02412-37 (Other: DGS, Ministry of Health)
Record Dates: First submitted 2021-06-16; First posted 2021-07-02 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stomach Neoplasms; Gastric Neoplasms; Helicobacter Pylori
Keywords: Helicobacter Pylori; Gastric cancer; Prevalence; French West-Indies
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained for extraction of DNA from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Helicobacter Pylori detection: Systematic biopsies of the tumor and the gastric cavity will be performed during the initial fibroscopy in accordance with the recommendations of the French Society of Digestive Endoscopy (SFED).
  Interventions: Biological: Helicobacter Pylori detection

INTERVENTIONS:
Biological: Helicobacter Pylori detection — Biopsies will be sent to the referral anatomopathology laboratory. The search for Helicobacter pylori will be performed by immunohistochemistry. An additional blood sample for serological testing will be taken during the initial workup.
  Additional data will be collected through a questionnaire.

SUMMARY:
Estimating the prevalence of Helicobacter Pylori infection in newly diagnosed stomach cancers in the West-Indies will help to understand the epidemiology of this cancer, which is over-incident in the West Indies compared to France. In addition, the constitution of a biobank (tumor tissues, healthy tissues and serum) will allow to set up in a second time etiological studies to identify other risk factors in particular in connection with the exposure to environmental pollutants to adapt the prevention measures.

DETAILED DESCRIPTION:
In the Antilles-Guyana, gastric cancer affects approximately 80 men and women each year in Guadeloupe and Martinique, and 20 in French Guiana. It is more frequent than in France and represents 4.5% of cancers in men in Martinique, 5.3% in Guadeloupe and 5.7% in French Guyana. It is the 3rd most common cancer site in men in Guadeloupe and Martinique, and the 4th in French Guiana. In women, it is the 3rd most frequent cancer in Martinique and the 4th in Guadeloupe, whereas it is less frequent in French Guiana.

Studies are needed to estimate this prevalence in the general population and in cancer patients. The prevalence of Helicobacter pylori infection is not well known in the general population in the Caribbean and when gastric cancer is diagnosed, the bacterium is rarely tested.

Dietary habits in our regions are characterized by a high consumption of salt (salted), meat and smoked fish. These dietary habits, common to some Southeast Asian countries, could partly explain the high incidence of stomach cancer observed. But environmental risk factors could also be involved.

Patients referred to gastroenterology with a suspected endoscopic diagnosis of gastric cancer will be offered to participate in the study after the fibroscopy has been performed and their consent will be obtained for the use of diagnostic specimen remains for research purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years of age, residing for at least 6 months in Martinique, with a primary diagnosis of gastric cancer
2. Patient having read the information note and having signed the consent to participate in the study
3. Patient with social security coverage

Exclusion Criteria:

1. Refusal to participate
2. Patient who could not answer the questionnaires
3. Patient not affiliated to a social security system
4. Patient not fluent in French
5. Patient under legal protection (legal protection, guardianship, curators, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients (with a suspected endoscopic diagnosis of gastric cancer) will be selected either at the Martinique University Hospital or at the Sainte-Marie clinic during consultations or hospitalizations.
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Estimation of the prevalence of Helicobacter pylori | At baseline
  Helicobacter Pylori has detected by immunohistochemistry in the stomach of patients with gastric cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisse JOACHIM-CONTARET, Principal Investigator — CHU Martinique
Locations (1):
- CHU Martinique, Fort-de-France, Martinique